CLINICAL TRIAL: NCT06289478
Title: Efficacy and Safety of Retrograde Intraarticular Injection Via Drain Tube, Topical Soaking of Tranexamic Acid (TXA), or Placebo in Elderly Patients With Femoral Neck Fractures Undergoing Bipolar Hemiarthroplasty
Brief Title: Efficacy and Safety of Retrograde Intraarticular Injection, Topical Soaking of Tranexamic Acid (TXA), or Placebo in Femoral Neck Fractured Patients Undergoing Cementless Bipolar Hemiarthroplasty
Acronym: TXA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Kanyakorn Riewruja, Doctor, King Chulalongkorn Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0151/67
Record Dates: First submitted 2024-02-25; First posted 2024-03-04 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Femoral Neck Fracture
Keywords: tranexamic acid; femoral neck fracture; bipolar hemiarthroplasty; topical; blood transfusion
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Retrograde Intraarticular Injection via Drain Tube (Experimental): Tranexamic acid will be injected retrograde to the joint via drain tube after surgical wound closure
  Interventions: Drug: Topical tranexamic acid administration
- Topical Soaking of Tranexamic Acid (Experimental): Tranexamic acid will be placed to soak the intramedullary canal of the femur and surgical area after sheath closure for 5 minutes and completely remove by sunction
  Interventions: Drug: Topical tranexamic acid administration
- Standard procedure (placebo) (Placebo Comparator): Standard wound irrigation
  Interventions: Drug: Topical tranexamic acid administration

INTERVENTIONS:
Drug: Topical tranexamic acid administration — Tranexamic acid will be topically administered in intervention groups

SUMMARY:
The goal of this Randomized controlled trial is to evaluate in household ambulatory, elderly patients sustaining femoral neck fracture who are subjected to be treat with cementless bipolar hemiarthroplasty. The main questions it aims to answer are:

* The efficacy in reducing blood transfusion for topical tranexamic acid administration
* The safety of tranexemic acid, topically used

As having undergone bipolar hemiarthroplasty surgery, participants will either receive retrograde intraarticular tranexamic acid injection via drain tube, or topical soaking administration.

Researchers will compare, with standard procedure (procedure), whether topically administered tranexamic acid would reduce rate of blood transfusion.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients (age > 60 years)
* Femoral neck fractures from low energy mechanism
* Household ambulator
* Undergoing cementless bipolar hemiarthroplasty at KCMH
* Informed consent

Exclusion Criteria:

* Allergy to TXA
* History of VTE
* History of hip surgery, pathological fracture, hip infection
* Congenital or acquired coagulopathy
* Hb < 10 g/dL or Platelet < 140,000

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Rate of blood transfusion | 2 years, or until complete enrollment
  Proportion of patients received blood transfusion divided by total number of patient in a group

SECONDARY OUTCOMES:
Volume of blood transfusion | 2 years, or until complete enrollment
  total volume of blood transfusion per each patient
Calculated blood loss | 2 years, or until complete enrollment
  Calculating using Nadler and Goss formula
Any adverse events | 2 years, or until complete enrollment
  Adverse events include wound complication, deep vein thrombosis, pulmonary embolism, and other complication
In-hospital mortality | During admission period
  In-hospital mortality

CONTACTS AND LOCATIONS:
Locations (2):
- Thailand (2):
  - Faculty of Medicine, King Chulalongkorn Memorial Hospital, Bangkok
  - Faculty of Medicine, Bangkok

IPD SHARING:
Plan to Share IPD: Undecided